CLINICAL TRIAL: NCT06019052
Title: Testing New Diagnostic Technology Classes for TB (DriveDx4TB)
Brief Title: Evaluating Next Generation LAM Assays and Molecular Diagnostics (POC and Near POC) for the Diagnosis of TB Among People With Presumptive TB: a Prospective Multicentre Diagnostic Accuracy Study
Acronym: DriveDx4TB
Status: Not yet recruiting | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: TB051
Record Dates: First submitted 2023-08-10; First posted 2023-08-31 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis
Keywords: TB; Diagnostics; HIV; Diagnostic accuracy study; Alternative samples; Point of care (POC); Near POC; Molecular diagnostic (MDx) platforms; Urine LAM
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This prospective multicentre study is planned to evaluate the next generation LAM assays and molecular diagnostics (POC and near POC) among people with presumptive Tuberculosis. The DriveDx4TB study aims to generate evidence needed to accelerate the introduction of three new classes of TB diagnostics, complemented by alternative sampling for use at primary healthcare and community settings. To this end, the study will leverage the accelerated innovation spurred by the COVID-19 pandemic, particularly the rapid development of swab-based sampling and molecular diagnostic (MDx) platforms.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a major global health problem owing to high rates of morbidity and mortality; the 2022 Global TB Report estimates that approximately 10.6 million individuals fell ill with TB in 2021, however on account of existing programme inefficiencies and compounded by the effects of COVID-19, 4.1 million people with TB went undiagnosed. Access to diagnostics remains a significant barrier to TB care, further exacerbated by COVID-19; the consequence of delayed diagnoses and subsequent treatment has resulted in increased TB deaths (1.4M deaths in 2021 - levels last seen in 2017). In addition, a reliance on sputum-based testing has limited case detection efforts, particularly among individuals with paucibacillary disease (e.g., people living with HIV [PLHIV] and children) and those investigated earlier in their TB disease progression, where sputum production is inherently difficult. New fit-for-purpose diagnostics are thus urgently needed to recover lost ground and to bring testing closer to patients and address current sampling limitations.

The DriveDx4TB project aims to generate evidence needed to accelerate the introduction of three new classes of TB diagnostics, complemented by alternative sampling for use at primary healthcare and community settings. To this end, the study will leverage the accelerated innovation spurred by the COVID-19 pandemic, particularly the rapid development of swab-based sampling and molecular diagnostic (MDx) platforms.

The project will independently evaluate three technology classes:

1. 3rd Generation urine LAM
2. Point-of-care (POC) MDx using tongue swabs
3. Near POC MDx using tongue swabs or sputum

The data gathered from this study will support in-country decision-making for the uptake of new TB diagnostics, and will form part of evidence reviewed by the WHO for policy development or prequalification (PQ) processes.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years), with presumptive pulmonary TB i.e., self-reporting cough ≥2 weeks and ≥1 other symptom typical of pulmonary TB*
* Willing to provide written informed consent
* Willing to provide sputum, and other samples (tongue swabs, urine)
* Willingness to have a telephonic follow-up call 2-3 months post-enrolment
* Documented HIV status and CD4 count within last 6 months, or if unavailable, then willing to undergo testing
* fever, night sweats or unintended weight-loss

Exclusion Criteria:

* Participants currently on anti-TB treatment *
* Any anti-TB treatment or antibiotics not specifically used for TB treatment, but which have anti-TB activity, e.g., fluoroquinolones given for respiratory tract infection within 60 days prior to enrolment
* Any tuberculosis preventive therapy (TPT) within 6 months prior to enrolment
* Participants who have conditions or circumstances that preclude their participation, based on the judgement of the site investigator
* Unable to produce at least 3ml of sputum * Participants starting anti-TB treatment at the time of enrolment will not be excluded from the study provided that all study specimens are collected before starting the 3rd dose of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 1800 Adult (≥18 years), with presumptive pulmonary TB i.e., self-reporting cough ≥2 weeks and ≥1 other symptom typical of pulmonary TB* will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1890 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
1.1 | February 2024 to August 2025
  Determination of the diagnostic accuracy of POC index tests using urine samples for TB detection among adults with presumptive pulmonary TB using as reference standards MRS, eMRS, and CRS. Point estimates (with 95% confidence intervals) of sensitivity, specificity, balanced accuracy, diagnostic odds ratio (DOR), positive and negative predictive values (PPV and NPV) for POC index tests using the defined MRS, eMRS and CRS as reference standards. Point estimates of sensitivity and specificity will be calculated based on the definitions reported in protocol, with 95% confidence intervals calculated using Wilson's score method.
  The efficacy analyses will be performed on the PP population. Additional subgroup analyses of the primary endpoints will be performed as per SAP.
1.2 | February 2024 to August 2025
  Determination of the diagnostic accuracy of near POC MDx index tests using tongue swabs for TB detection among adults with presumptive pulmonary TB using as reference standards MRS, eMRS and CRS. Point estimates (with 95% confidence intervals) of sensitivity, specificity, balanced accuracy, DOR, PPV and NPV for near POC MDx index tests, using the defined MRS, eMRS and CRS as reference standards. Point estimates of sensitivity and specificity will be calculated based on the definitions reported in protocol with 95% confidence intervals calculated using Wilson's score method.
  The efficacy analyses will be performed on the PP population. Additional subgroup analyses of the primary endpoints will be performed as per SAP.
1.3 | February 2024 to August 2025
  Determination of the diagnostic accuracy of low complexity NAAT index tests using tongue swabs or sputum for TB detection among adults with presumptive pulmonary TB using as reference standards MRS, eMRS and CRS.Point estimates (with 95% confidence intervals) of sensitivity, specificity, balanced accuracy, DOR, PPV and NPV for low complexity index tests, using the defined MRS, eMRS and CRS as reference standards.Point estimates of sensitivity and specificity will be calculated based on the definitions reported in protocol with 95% confidence intervals calculated using Wilson's score method.
  The efficacy analyses will be performed on the PP population. Additional subgroup analyses of the primary endpoints will be performed as per SAP.

SECONDARY OUTCOMES:
2.1 | February 2024 to August 2025
  Comparison of the diagnostic accuracy between index tests and a comparator test or combinations belonging to the same technology class (POC, near POC MDx or low complexity NAAT), for TB detection among adults with presumptive pulmonary TB. Difference between the point estimates (with 95% confidence intervals) of sensitivity and specificity for each index test and its relative comparator test, using MRS, eMRS and CRS as reference standards. Point estimates of sensitivity and specificity will be calculated based on the definitions reported in protocol with 95% confidence intervals calculated using Wilson's score method.
  The efficacy analyses will be performed on the PP population. Additional subgroup analyses of the primary endpoints will be performed as per SAP.
2.2 | February 2024 to August 2025
  Determination of the diagnostic accuracy of POC index tests using urine samples, of near POC MDx index tests using tongues swabs, and of near POC MDx index tests using tongue swabs or sputum for TB detection among adults with presumptive pulmonary TB and HIV infection using MRS, eMRS and CRS. Point estimates (with 95% confidence intervals) of sensitivity, specificity, balanced accuracy, DOR, PPV and NPV for POC index tests using urine samples, near POC MDx index tests using tongues swabs, and low complexity NAAT index tests using tongue swabs or sputum, in the TB and HIV co-infection subgroup using MRS, eMRS and CRS as reference standards.
2.3 | February 2024 to August 2025
  Evaluation of the usability of POC, of near POC MDx and of low complexity NAAT index tests in a real-world setting. Usability of each index test (3rd generation LAM, near POC MDx and low complexity NAAT) measured by the operators' ability to understand the test instructions, workflow and results interpretation.

IPD SHARING:
Plan to Share IPD: No